CLINICAL TRIAL: NCT03218670
Title: Your Health in On Click : Risk Behavior Among College Students
Brief Title: Your Health in On Click
Acronym: TS1C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marie-Pierre TAVOLACCI (Other)
Responsible Party: Sponsor-Investigator, Marie-Pierre TAVOLACCI, Doctor, University Hospital, Rouen
Organization: University Hospital, Rouen (Other)
Other Study IDs: 2016/307/OB
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: College Student Drinking; Eating Disorder; Stress, Psychological; Burn Out Syndrome; Cigarette Smoking; Hyperactivity; Health Behavior; Impulsive Behavior
MeSH Terms: conditions — Alcohol Drinking in College; Feeding and Eating Disorders; Stress, Psychological; Burnout, Psychological; Cigarette Smoking; Spasm; Health Behavior; Impulsive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A health education program was provided to higher education students aged between 18 and 25 years. Students were recruited either by posters and leaflets on campus, or during their mandatory medical survey at the University Medical Department. The objectives are to assess health behavior risk among college student : e.g eating disorders, binge drinking, electronic cigarettes and also stress, burnout

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years
* College students

Exclusion Criteria:

* No college students

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: College students in France
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2009-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of binge drinking, eating disorders, burn out and other risk behaviors among college students | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Tavolacci, Rouen, France

IPD SHARING:
Plan to Share IPD: No